CLINICAL TRIAL: NCT05562284
Title: Safety and Efficacy of the Visual Field Improvement After Selective Intra-arterial Thrombolysis for Central Retinal Artery Occlusion
Brief Title: Safety and Efficacy After Selective Intra-arterial Thrombolysis for Central Retinal Artery Occlusion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Ping Fei, Associate professor, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XHEC-C-2022-056
Record Dates: First submitted 2022-08-29; First posted 2022-09-30 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Central Retinal Artery Occlusion
Keywords: central retinal artery occlusion; intra-arterial thrombolysis; visual field
MeSH Terms: conditions — Retinal Artery Occlusion | interventions — Conservative Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IAT combined with conservative therapies (Experimental): IAT (Drug: 50 mg Alteplase)+conservative treatments
  Interventions: Procedure: intra-arterial thrombolysis; Other: conservative treatments
- Conservative therapies (Other): conservative treatments including traditional ones and hyperbaric oxygen therapy
  Interventions: Other: conservative treatments

INTERVENTIONS:
Procedure: intra-arterial thrombolysis — IAT introduces rt-PA directly into the ophthalmic circulation by super-selective microcatheterization.
  Arms: IAT combined with conservative therapies
Other: conservative treatments — conservative treatments

SUMMARY:
Central retinal artery occlusion (CRAO) is an ophthalmic emergency which leads to devastating visual function defects and poor prognosis. Though traditional conservative treatments are widely used, none of them is proved to be effective. A number of meta-analyses and observational studies indicate intravenous thrombolysis to be beneficial in CRAO. Selective intra-arterial thrombolysis (IAT) introducing rt-PA directly into the ophthalmic circulation by super-selective microcatheterization may reduce the complications such as intracranial and systemic hemorrhage.The residual visual field is significant for patients with CRAO who have poor central visual acuity. Thus, it is clinically significant to study the changes in visual fields in eyes with CRAO.

DETAILED DESCRIPTION:
Central retinal artery occlusion (CRAO) is an ophthalmic emergency which leads to devastating visual function defects and poor prognosis. Though traditional conservative treatments are widely used, none of them is proved to be effective. The respective responses of brain and retinal tissues to acute ischemia share many features is the rationale for therapeutic thrombolysis in CRAO. Intravenous thrombolysis (IVT) has been a therapeutic choice for CRAO since the 1960s, and in the United States, tPA is currently administered in 5.8% of patients admitted with CRAO. A number of meta-analyses and observational studies indicate intravenous thrombolysis to be beneficial in CRAO. Selective intra-arterial thrombolysis (IAT) introducing rt-PA directly into the ophthalmic circulation by super-selective microcatheterization which has the advantage of reducing the dose of rt-PA reaching the systemic circulation. Thus, IAT may reduce the complications such as intracranial and systemic hemorrhage. The residual visual field is significant for patients with CRAO who have poor central visual acuity. Thus, it is clinically significant to study the changes in visual fields in eyes with CRAO. Sequential evaluation by Humphrey perimetry will evaluate the temporal changes before and after IAT or conservative therapies. Our study will enroll patients within 7 days of symptom onset and aims at evaluating the safety of IAT and comparing the improvement of the VFDs between conservative treatments and IAT combined with conservative treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Non-arteritic CRAO with symptom duration ≤7d
2. Age from 18 years old between 80 years old
3. Qualified systemic conditions, well-controlled blood pressure, well-controlled blood glucose, qualified liver and kidney function, no allergic history to contrast agent or rt-PA,
4. Meet the inclusion of HBOT

Exclusion Criteria:

* Ocular factor or disease

  1. Branch retinal artery occlusion
  2. Combined retinal vein occlusion
  3. Suspicious ocular ischemic syndrome, such as ophthalmic artery occlusion or carotid artery occlusion
  4. Existed retinal problems decreasing visual function, such as macular disease, severe nonproliferative or proliferative diabetic retinopathy, severe cataract or glaucoma
  5. Central retinal artery occlusion from iatrogenic cause
  6. History of thrombolysis for CRAO or CRVO
* Systemic factors restricting thrombolysis

  1. Uncontrolled hypertension (systolic blood pressure > 180mmHg ); Uncontrolled hyperglycemia (fasting blood glucose > 9mmol/L);
  2. Coagulation disorder
  3. History of intracranial hemorrhage, heart attack, cerebral infarction, or intracranial surgery within 3 mo
  4. Current antithrombotic treatment
  5. History of allergic reaction to contrast agent or rt-PA

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Change of the visual field index as mean deviation (MD) examed by Humphrey visual field analyzer at 3 months | 90 days
  Change of the mean deviation
Change of the visual field index as visual field index (VFI) examed by Humphrey visual field analyzer at 3 months | 90 days
  Change of the visual field index

SECONDARY OUTCOMES:
Change of Best corrected visual acuity (BCVA) at 3 months | 90 days
  best corrected visual acuity of logarithm of the minimum angle of resolution
Adverse reactions at 1 month | 30 days
  Death, symptomatic or asymptomatic intracranial hemorrhage, intraocular hemorrhage

CONTACTS AND LOCATIONS:
Overall Officials: Ping Fei, MD#PhD, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Xinhua Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
protocols
Supporting Information: Study Protocol
Time Frame: 90 days after the interventions
Access Criteria: if required propriately